CLINICAL TRIAL: NCT04355975
Title: Clinical Outcomes After Acute Pulmonary Embolism - The Bern Acute Pulmonary Embolism Registry
Brief Title: Clinical Outcomes After Acute Pulmonary Embolism
Acronym: ERASE PE
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 4303 - 2019-02042
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Medical Therapy / Anticoagulation
- Systemic Lysis
- Interventional Therapy for PE
- Surgical Embolectomy

SUMMARY:
To investigate safety and effectiveness of PE treatment according to the decision of the multi-disciplinary pulmonary embolism response team (PERT) and to define and optimize treatment indications, institutional algorithms and interventional techniques for PE.

DETAILED DESCRIPTION:
This single-center cohort study is designed to retrospectively and prospectively collect treatment and outcome data related to patients with PE and after activation of the PERT. Treatment information and outcomes after advanced treatment modalities, including systemic thrombolysis, catheter directed thrombolysis and surgical embolectomy, will be collected.

Retrospective patient data will consist of treatment and health related outcomes of consecutive patients treated for acute and chronic PE between October 2017 and April 2020 (to assess the learning curve of the PERT) and of patients receiving surgical embolectomy between January 2001 and April 2020. The retrospective data will be derived from the local institutional dataset and will be transferred to the study database. Prospective patients will be included after May 2020.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with pulmonary embolism matching the criteria for treatment according to the decision of the PERT.
* Written informed consent

Exclusion Criteria:

* High probability of non-adherence to the follow up requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with Acute PE
  * Patients developing CTEPH
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital death | 30 days

SECONDARY OUTCOMES:
Peri-procedural adverse events | 30 days
Recurrent VTE during follow-up | up to 5 years
Respiratory and functional deterioration after treatment | 6 months
Development of chronic thromboembolic pulmonary hypertension (CTEPH) | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Stortecky, MD, Principal Investigator — Department of Cardiology, Bern University Hospital, University of Bern, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital Bern - Inselspital, Bern, Canton of Bern
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Draxler DF, Johannes JK, Nakase M, Heg D, Dobner S, Turovskij E, Furholz M, Haner J, Lanz J, Pilgrim T, Hunziker L, Praz F, Raber L, Rohla M, Siontis GCM, Susuri-Pfammatter N, Windecker S, Stortecky S. Clinical Outcomes in Patients With Acute Pulmonary Embolism Undergoing Ultrasound-Assisted Catheter-Directed Thrombolysis. J Am Heart Assoc. 2025 May 6;14(9):e035916. doi: 10.1161/JAHA.124.035916. Epub 2025 Apr 25. PMID 40281654